CLINICAL TRIAL: NCT01438268
Title: Expedited Discharge of Patients Undergoing Pedicled TRAM Flap Breast Reconstruction Procedure in Ambulatory Surgical Facility: Quality of Recovery Outcomes
Brief Title: TRAM Procedure in Ambulatory Surgical Facility: Quality of Recovery Outcomes
Acronym: TRAM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Women's College Hospital (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2010-0050-E
Record Dates: First submitted 2011-06-21; First posted 2011-09-22 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Breast Diseases
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Reconstructive breast cancer patients: Patients having unilateral, bilateral immediate or delayed TRAM flaps who are discharged 18 hours postoperatively

SUMMARY:
Specific Aim: To assess the quality of recovery of patients following early discharge (18 hrs) after pedicled TRAM flap breast reconstruction. Quality of recovery will be assessed using a 27-item validated questionnaire, QoR-27 at discharge, and on Post Operative Days (POD) 2, 4 and 7. In addition a 100 mm Visual Analog Score (VAS) for Pain will be completed on discharge from the recovery room, discharge from hospital and on POD 2, 4 and 7.

Clinical Relevance: Postoperative recovery is a complex process related to various outcomes such as physiological endpoints, incidence of adverse events and change in psychological status. Previous studies of recovery after surgery and anesthesia have focused primarily on the physiological endpoints and the incidence of adverse events. Much of the work has occurred in specialties dealing with chronic disease states such as cancer, rheumatology and musculoskeletal disorders. There is clearly a need to focus on recovery outcome measures in the ambulatory population for postoperative recovery. Here the investigators propose to measure postoperative recovery outcomes within the first week following a TRAM flap reconstructive procedure using a validated postoperative quality of recovery instrument (QoR-27) and a 100 mm VAS for pain.

DETAILED DESCRIPTION:
Women's College Hospital is the first and only independent ambulatory care hospital in Ontario, and the only hospital in Ontario with a primary focus on women's health. Patients undergoing breast reconstruction following breast cancer at our institution are now undergoing expedited discharge at 18 hrs postoperatively. To facilitate next day discharge, a multidisciplinary group was formed to determine the best evidence for perioperative care to ensure patient safety and excellent postoperative recovery. Minimizing length of stay has obvious cost savings for hospitals, but for patients the advantages include minimizing exposure to hospital-acquired infections and an earlier return to their more familiar home environment. The need to balance the advantage of early discharge to patient complications, however, must be addressed. As other hospitals across the country face the same length of stay constraints as has been our experience, this study will provide important data on the quality of recovery of patients undergoing early discharge following breast reconstructive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing any type of TRAM flap
* Age<75 yrs
* Non-smoker

Exclusion Criteria:

* History of chronic pain or psychiatric disturbance
* History of chronic use of opioid medications
* Allergy to local anesthesia or opioid medication
* Inability to communicate in English
* BMI>35

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Reconstructive breast cancer patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-08 (Actual); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the quality of recovery at discharge as assessed by the QoR27 | On average between 18 and 24 hours postoperatively
  The patient will be met with by the study coordinator, just before discharge to administer the Quality of Recovery Questionnaire (QoR27)
The primary outcome measure is the quality of recovery post operatively, as assessed by the QoR27 | on average between 48-72 hours postoperatively
  The patient will be contacted by the study coordinator, 2 days following their surgery to administer the Quality of Recovery Questionnaire (QoR27)
The primary outcome measure is the quality of recovery at discharge as assessed by the QoR27 | On average 72-96 hours post operatively
  The patient will be contacted by the study coordinator, 4 days following their surgery to administer the Quality of Recovery Questionnaire (QoR27)
The primary outcome measure is the quality of recovery post operatively as assessed by the QoR27 | On average 7-8 days postoperatively
  The patient will be contacted by the study coordinator, 7 days following their surgery to administer the Quality of Recovery Questionnaire (QoR27)

SECONDARY OUTCOMES:
The secondary outcome measure is the quality of recovery as assessed by the VAS pain score | This outcome will be done at the exact same time as the measurements of Quality of Recovery listed above
  These scores will be compared

CONTACTS AND LOCATIONS:
Overall Officials: John L Semple, MD, MSc, FRCSC, FACS, Principal Investigator — Women's College Hospital; Pamela J Morgan, MD, CCFP, FRCPC, Study Director — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada